CLINICAL TRIAL: NCT04655573
Title: A Pilot Study of a Micro-Organosphere Drug Screen Platform to Lead Care in Advanced Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: requested by sponsor
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107118
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Advanced Breast Cancer
Keywords: Patient derived micro-organospheres (PDMO); Chemotherapy; Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Patient derived tumor specimens that are cultured into patient-derived micro-organospheres (PDMO) for patients with ABC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient Derived Micro-Organospheres (PDMO): Subjects will undergo image-guided biopsy as a standard of care clinical biopsy from which extra tissue is taken for research purposes. Following the biopsy, a PDMO will be generated and they will receive a chemotherapy regimen as determined by their treating physician. PDMO are successfully generated, and the patient begins treatment with a hemotherapy backbone. A patient will be considered evaluable if pathology results are available from the biopsy.
  Interventions: Procedure: Breast Cancer Tumor Resection

INTERVENTIONS:
Procedure: Breast Cancer Tumor Resection — Patients with ABC will be receiving a biopsy, and a PDMO from the patient's biopsies will be generated from it. It is a model correlating clinical response with PDMO sensitivity to the most common forms of chemotherapy used in advanced breast cancer care.

SUMMARY:
The purpose of this study is to assess the feasibility of generating patient derived micro-organospheres (PDMO) from patients with advanced breast cancer to determine sensitivity to the most common forms of chemotherapy used in advanced breast cancer care.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of generating sufficient patient derived micro-organospheres (PDMO) from a biopsy of a patient's advanced breast cancer to determine sensitivity to the most common forms of chemotherapy used in advanced breast cancer care. While subjects are on study, they will first receive a standard of care clinical biopsy from which extra tissue is taken for research purposes. Following the biopsy, a PDMO will be generated and they will receive a chemotherapy regimen as determined by their treating physician. This study aims to enroll 15 patients. Of this 15 patient cohort we aim to enroll 5 patients with estrogen receptor positive (ER+)/human epidermal growth factor receptor 2 negative (HER2-) disease, 5 patients with ER+/HER2+ or ER-/HER2+ disease, and 5 patients with ER-/HER2- (TNBC) disease. There are risks to having biopsies and blood draws that may include moderate bleeding and pain at the biopsy site.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Female ages 18 or older.
3. Have measurable disease ≥ 2 cm defined by RECIST version 1.1.
4. Amenable to standard of care biopsy with co-consent to the Duke BioRepository & Precision Pathology Center (BRPC) protocol (Pro00035974) to collect extra biopsy tissue for research or willing to provide extra tissue other than standard of care without co-consent to BRPC.
5. Evidence of advanced cancer of the breast that is surgically unresectable with pathology confirming ER, PR, and HER2 status. NOTE: patients may enroll prior to receiving clinical biopsy results based on historical pathology results.
6. Patient is eligible for chemotherapy as monotherapy or in combination with single-agent anti HER2 Therapy.

   * ER+/PR+/HER2-, must have progressed or be intolerant to CDK 4/6 inhibitor and/or endocrine therapy unless CDK 4/6 inhibitor is not able to be provided per the clinician's discretion endocrine therapy and CDK 4/6 inhibitor
   * ER+/PR+/HER2+ or ER-/PR-HER2+, must have progressed or be intolerant to ≥ 2 lines of anti-HER2 therapy and be considered for mono-chemotherapy with trastuzumab and/or anti-HER2 tyrosine kinase inhibitor
   * ER-/PR-HER2-, PD-L1- and/or TMB <10 may may be considered for first line of treatment
7. Treating physician is planning to treat breast cancer in the advanced setting with a chemotherapy backbone. This study excludes patients who will receive an antibody-drug conjugate as their proposed treatment.
8. Impending visceral crisis is allowed only if the patient can have a biopsy prior to starting systemic mono-chemotherapy
9. ECOG performance status of 0, 1, or 2.
10. Any metastatic site that is ≥ 2cm and amenable to core needle biopsy. Patients with brain metastases are allowed and MOS may be generated from a resected breast cancer brain metastasis

Exclusion Criteria:

1. Actively requiring systemic antibiotics.
2. Clinically significant cardiac disease, including unstable angina or acute myocardial infarction within 6 months of enrollment.
3. Leptomeningeal disease
4. Pregnant women.
5. Enrolling on an investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with advanced breast cancer
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with successful generation of PDMO from the patient's biopsy | 10 days of biopsy
  The PDMO establishment will be monitored and success will be defined as the formation of 3D organoid structures in at least 80% of droplets in each well, in 20 randomly sampled wells per PDMO model, within 7 days. With an anticipated generation of 90% we anticipate being able to generate 13 PDMO from the first 15 patients to perform a drug screen within 10 days of biopsy. The exact 90% lower confidence bound (LCB) will be computed for the proportion of patients with successful generation of PDMO and completed drug screen within 10 days. For the first 6 patients, if at least 5 PDMO can be generated and screened on 6 patients' samples the procedure will be deemed feasible. With 6 patients studied the exact 90% LCB assuming 5 successful cases is 0.71. We would thus be 90% confident that the success rate of this strategy is at least 71%.

SECONDARY OUTCOMES:
Association between specific chemotherapy sensitivity in PDMO to clinical outcome of patient | End of study (up to 2 years)
  For the 15 evaluable patients, the MODEL ABC platform will be used to assess sensitivity to chemotherapy and generate a prediction model for correlation with patient data. For each sample, two primary outcomes will be collected: i) PDMO drug sensitivity data, and ii) the patient's clinical outcome (PFS). Treating PDMO with 10 chemotherapy single agents at 10 drug concentrations each will generate drug sensitivity data. For all 15 samples, PDMO sensitivity to each concentration of each drug will be used alongside the 15 clinical responses (PFS) to develop a predictor of PFS by correlating drug response data to clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dent, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No